CLINICAL TRIAL: NCT01095666
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 3 Trial to Evaluate the Safety and Efficacy of Dapagliflozin in Combination With Metformin in Asian Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin Alone
Brief Title: A Phase III Study of BMS-512148 (Dapagliflozin) in Asian Patients With Type 2 Diabetes Who Are Not Well Controlled on Metformin Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: AstraZeneca, Bristol-Myers Squibb (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB102-055
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Metformin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental)
  Interventions: Drug: Dapagliflozin; Drug: Metformin; Drug: Dapagliflozin Placebo; Drug: Pioglitazone
- Group 2 (Experimental)
  Interventions: Drug: Dapagliflozin; Drug: Metformin; Drug: Dapagliflozin Placebo; Drug: Pioglitazone
- Group 3 (Experimental)
  Interventions: Drug: Metformin; Drug: Dapagliflozin Placebo; Drug: Pioglitazone

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 5 mg, Once daily, 24 weeks
  Other Names: BMS-512148
  Arms: Group 1
Drug: Dapagliflozin — Tablets, Oral, 10 mg, Once daily, 24 weeks
  Other Names: BMS-512148
  Arms: Group 2
Drug: Metformin — Tablets, Oral, 1500-3000 mg, Twice daily, 24 weeks
  Other Names: Glucophage®
Drug: Dapagliflozin Placebo — Tablets, Oral, 0 mg, Once daily, 24 weeks
Drug: Pioglitazone — Tablets, Oral, 15-45 mg (as needed for rescue based on protocol specific criteria), Up to 20 weeks

SUMMARY:
The purpose of this clinical research study is to learn if BMS-512148 (Dapagliflozin) can help reduce the blood sugar levels in Asian patients with Type 2 Diabetes who are not well controlled on metformin alone. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 to 77 years old, with type 2 diabetes and with inadequate glycemic control
* Drug naive or treated with anti-diabetic medication for < 24 weeks
* C-peptide ≥ 1.0 ng/mL
* Body Mass Index ≤ 45.0 kg/m²

Exclusion Criteria:

* AST and/or ALT > 3 times ULN
* Serum total bilirubin > 2 mg/dL
* Serum creatinine ≥ 1.50 mg/dL for men or ≥ 1.40 mg/dL for women
* Creatine kinase ≥ 3 times ULN
* Symptoms of severely uncontrolled diabetes
* Currently unstable or serious cardiovascular, renal, hepatic, hematological, oncological, endocrine, psychiatric, or rheumatic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1484 (Actual)
Dates: Start 2010-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- China (16):
  - Local Institution, Hefei, Anhui
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Chongqing, Chongqing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Haerbin, Heilongjiang
  - Local Institution, Changsha, Hunan
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Wuxi, Jiangsu
  - Local Institution, Changchun, Jilin
  - Local Institution, Shenyang, Liaoning
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Chongqing, Sichuan
  - Local Institution, Tianjin, Tianjin Municipality
  - Local Institution, Hangzhou, Zhejiang
  - Local Institution, Xi'an
- India (5):
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Indore, Madhya Pradesh
  - Local Institution, Bangalore
  - Local Institution, Jaipur
  - Local Institution, Vellore, Tamilnadu
- South Korea (3):
  - Local Institution, Seoul, Nowon-Gu
  - Local Institution, Busan
  - Local Institution, Seoul

REFERENCES:
- See also: Publication — https://www.ncbi.nlm.nih.gov/pubmed/26589253

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 1484 patients enrolled, 554 completed a qualification period. Of these 554 patients, 444 were randomized and received treatment. Of these 444 participants, 409 completed the double-blind treatment period
Period: Overall Study
Arm/Group | Placebo + Metformin | Dapagliflozin 5 mg + Metformin | Dapagliflozin 10 mg + Metformin
Started | 145 | 147 | 152
Completed | 128 | 136 | 145
Not Completed | 17 | 11 | 7
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Adverse Event | 2 | 1 | 3
Not completed — Lost to Follow-up | 2 | 2 | 0
Not completed — Withdrawal by Subject | 6 | 6 | 1
Not completed — Non-compliance, not met criteria etc. | 7 | 2 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Metformin | Dapagliflozin 5 mg + Metformin | Dapagliflozin 10 mg + Metformin | Total
Number analyzed (Participants) | 145 | 147 | 152 | 444
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (9.20) | 53.1 (9.09) | 54.6 (9.54) | 53.8 (9.29)
Age, Customized [Number; unit: Participants]
  Yonger than 65 years | 129 | 132 | 126 | 387
  65 to younger than 75 years | 14 | 13 | 25 | 52
  75 years and older | 2 | 2 | 1 | 5
Sex/Gender, Customized [Number; unit: Participants]
  Male | 86 | 67 | 88 | 241
  Female | 59 | 80 | 64 | 203
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian Indian | 10 | 11 | 13 | 34
  Chinese | 126 | 127 | 129 | 382
  Korean | 9 | 9 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1C (HbA1c) at Week 24 (Last Observation Carried Forward [LOCF])
Description: HbA1c was measured as percent of hemoglobin by a central laboratory. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. HbA1c measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 4, 8, 12, 16, 20, and 24 in the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing HbA1c values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: % of hemoglobin
Arm/Group | Placebo + Metformin | Dapagliflozin 5 mg + Metformin | Dapagliflozin 10 mg + Metformin
Number analyzed (Participants) | 139 | 146 | 149
% of hemoglobin | -0.23 (0.0622) | -0.82 (0.0607) | -0.85 (0.0601)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Dapagliflozin 5 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Primary endpoints were tested at alpha=0.027 applying Dunnett's adjustment; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-0.76 to -0.42], Standard Error of Mean 0.0869
Statistical Analysis 2: Comparison: Placebo + Metformin vs Dapagliflozin 10 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Primary endpoints were tested at alpha=0.027 applying Dunnett's adjustment; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-0.79 to -0.45], Standard Error of Mean 0.0865

2. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Fasting plasma glucose was measured as milligrams per deciliter(mg/dL) by a central laboratory. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. FPG measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 1, 2, 4, 8, 12, 16, 20, and 24 in the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing FPG values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo + Metformin | Dapagliflozin 5 mg + Metformin | Dapagliflozin 10 mg + Metformin
Number analyzed (Participants) | 140 | 146 | 151
mg/dL | 0.5 (2.357) | -21.6 (2.308) | -26.6 (2.269)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Dapagliflozin 5 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -22.1, 95% CI 2-sided [-28.6 to -15.6], Standard Error of Mean 3.299
Statistical Analysis 2: Comparison: Placebo + Metformin vs Dapagliflozin 10 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -27.1, 95% CI 2-sided [-33.5 to -20.7], Standard Error of Mean 3.271

3. Secondary Outcome: Adjusted Mean Change From Baseline in 2-hour Post Meal Glucose (PMG) (mg/dL) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Post Meal Glucose was measured as milligrams per deciliter(mg/dL) by a central laboratory. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. PMG measurements were obtained on Day 1 and week 24 in the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing PMG values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo + Metformin | Dapagliflozin 5 mg + Metformin | Dapagliflozin 10 mg + Metformin
Number analyzed (Participants) | 117 | 117 | 124
mg/dL | -15.5 (4.1548) | -57.8 (4.1547) | -64.6 (4.0357)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Dapagliflozin 5 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -42.3, 95% CI 2-sided [-53.84 to -30.73], Standard Error of Mean 5.8758
Statistical Analysis 2: Comparison: Placebo + Metformin vs Dapagliflozin 10 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -49.1, 95% CI 2-sided [-60.53 to -37.74], Standard Error of Mean 5.7921

4. Secondary Outcome: Adjusted Mean Change From Baseline in Total Body Weight (kg) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Adjusted mean change from baseline in total body weight at Week 24 (or the last postbaseline measurement prior to Week 24 if no Week 24 assessment was available was determined. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Body weight measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 1, 2, 4, 8, 12, 16, 20, and 24 of the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing body weight values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo + Metformin | Dapagliflozin 5 mg + Metformin | Dapagliflozin 10 mg + Metformin
Number analyzed (Participants) | 141 | 147 | 151
kg | -0.74 (0.1975) | -1.84 (0.1935) | -2.56 (0.1909)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Dapagliflozin 5 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -1.10, 95% CI 2-sided [-1.65 to -0.56], Standard Error of Mean 0.2765
Statistical Analysis 2: Comparison: Placebo + Metformin vs Dapagliflozin 10 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -1.82, 95% CI 2-sided [-2.36 to -1.28], Standard Error of Mean 0.2747

5. Secondary Outcome: Participants Achieving a Therapeutic Glycemic Response (Hemoglobin A1c [HbA1C]) <7.0% at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Therapeutic glycemic response is defined as HbA1c <7.0%. Data after rescue medication was excluded from this analysis. HbA1c was measured as a percent of hemoglobin. Percentage of participants were estimated by modified logistic regression model, adjusted for baseline HbA1c.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing HbA1C values at Week 24 (LOCF)
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Metformin | Dapagliflozin 5 mg + Metformin | Dapagliflozin 10 mg + Metformin
Number analyzed (Participants) | 139 | 146 | 149
Percentage of Participants | 17.5 (3.136) [11.3 to 23.6] | 32.9 (3.667) [25.7 to 40.1] | 33.0 (3.528) [26.1 to 39.9]
Statistical Analysis 1: Comparison: Placebo + Metformin vs Dapagliflozin 5 mg + Metformin; Test type: Superiority or Other; p = 0.0010, Modified logistic regression — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Modified logistic regression model, adjusted for baseline HbA1c; Difference in percentage = 15.4, 95% CI 2-sided [6.2 to 24.7], Standard Error of Mean 4.702
Statistical Analysis 2: Comparison: Placebo + Metformin vs Dapagliflozin 10 mg + Metformin; Test type: Superiority or Other; p = 0.0007, Modified logistic regression — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Modified logistic regression model, adjusted for baseline HbA1c; Difference in percentage = 15.5, 95% CI 2-sided [6.5 to 24.5], Standard Error of Mean 4.594

ADVERSE EVENTS:
Time Frame: Onset on or after the first date of double-blind treatment and on or prior to the last day of double-blind treatment 24 weeks plus 4 days for non-serious adverse event; plus 30 days for serious adverse event.
Arm/Group | Placebo + Metformin | Dapagliflozin 5 mg + Metformin | Dapagliflozin 10 mg + Metformin
Serious Adverse Events (participants affected / at risk) | 6/145 | 3/147 | 3/152
Other Adverse Events (participants affected / at risk) | 34/145 | 43/147 | 42/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Metformin (N=145) | Dapagliflozin 5 mg + Metformin (N=147) | Dapagliflozin 10 mg + Metformin (N=152)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
JOINT INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
INFLAMMATORY PSEUDOTUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL BRIDGING (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Metformin (N=145) | Dapagliflozin 5 mg + Metformin (N=147) | Dapagliflozin 10 mg + Metformin (N=152)
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 16 (17) | 18 (18) | 18 (19)
URINARY TRACT INFECTION (Infections and infestations) | 7 (8) | 6 (6) | 10 (15)
NASOPHARYNGITIS (Infections and infestations) | 5 (5) | 9 (9) | 7 (7)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 14 (16) | 6 (6)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 8 (12) | 6 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No